CLINICAL TRIAL: NCT04553718
Title: Construct and Evaluate the Effectiveness of a Theory-based mHealth for Overweight and Obese Women --Develop Applications With Wearable Devices
Brief Title: Construct and Evaluate the Effectiveness of a Theory-based mHealth for Overweight and Obese Women During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, head of administration, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MackayMedical
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gestational Weight Gain; Physical Activity
Keywords: overweight; obese; pregnant women
MeSH Terms: conditions — Gestational Weight Gain; Motor Activity; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiemental group (Experimental): Experimental group was the mHealth app to improved their gestational weight gain and physical activity during pregnancy.
  Interventions: Other: experimental group
- control group (No Intervention): standard prenatal care and without mHealth app

INTERVENTIONS:
Other: experimental group — provide mHealth program, which has pregnant women using wearable device and app
  Arms: experiemental group

SUMMARY:
This study was to construct and develop an application (APP) based on social-cognitive theory for overweight and obese women during pregnancy.

DETAILED DESCRIPTION:
Our program used and evaluated the mHealth program, which has pregnant women using APP and wearable devices to help prevent excessive gestational weight gain, and it continued to promote physical activity for overweight and obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

pregnant women--who have had, for 8-12 weeks, a pre-pregnancy body mass index of more than 25 kg/m2

Exclusion Criteria:

high risk pregnancy, such as pre-clampsia, pregnancy induced hypertension, preterm contraction

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Manage gestational weight gain | 4-6 week
  control excessive gestational weight gain

SECONDARY OUTCOMES:
Increase physical activity level | 4-6 week
  increase the scores of pregnancy of physical activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ching Fang Lee, PhD, Principal Investigator — Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No